CLINICAL TRIAL: NCT06621589
Title: The Effect of Nutritional Counseling on Anthropometry, Body Composition, Total Cholesterol, Blood Glucose, Uric Acid Levels, Attitude, and Behavior in Female Workers Wih Obesity at Adam Malik Hospital, Indonesia
Brief Title: Effect of Nutritional Counseling on Health Outcomes in Female Workers Wih Obesity at Adam Malik Hospital
Acronym: ECHO-OFEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RS H Adam Malik (Other)
Responsible Party: Principal Investigator, Hilna Khairunisa Shalihat, Head of Nutrition Unit, RS H Adam Malik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1084/KEPK/USU/2024
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: Nutritional Counseling; Obesity; Female Employees; Anthropometry; Body Composition; Lipid Profile; Uric Acid Levels; Blood Glucose; HbA1c; Quasi-Eksperimental Study; Adam Malik Hospital; Medan; Dietary Intervention
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: This study is a quasi-experimental design with a single group of participants receiving nutritional counseling. The participants will undergo pre- and post-intervention assessments to measure changes in health indicators, attitudes, and behaviors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutritional Counseling Group (Experimental): Participants in this arm will receive personalized nutritional counseling sessions aimed at improving their dietary habits, attitudes, and overall health outcomes. The counseling will take place over a 8-week period, and participants will undergo assessments before and after the intervention to evaluate changes in anthropometric measurements, body composition, and various health metrics.
  Interventions: Behavioral: Nutritional Counseling

INTERVENTIONS:
Behavioral: Nutritional Counseling — The intervention involves nutritional counseling aimed at improving dietary habits and overall health to participants. During the 2-month period, participants will receive guidance on nutrition, diet planning, and lifestyle changes tailored to their needs. Assessments of knowledge, attitudes, and health metrics will be conducted before and after the counseling sessions to measure the effectiveness of the intervention

SUMMARY:
The goal of this quasi-experimental study is to determine whether nutritional counseling can improve health outcomes in female workers with obesity at Adam Malik Hospital in Medan. Specifically, the study aims to assess the impact of nutritional counseling on participants; anthropometric measurements, body composition, total cholesterol, blood glucose, uric acid levels, as well as on attitudes, and behavioral changes.

The main questions it aims to answer are:

* What are the effects of nutritional counseling on anthropometric measurements, body composition, total cholesterol, blood glucose, uric acid levels?
* How does nutritional counseling affect attitudes toward healthy eating and changes in health behaviors?

Researchers will compare the health metrics of participants before and after receiving nutritional counseling to evaluate its effectiveness.

Participants will:

* Attend personalized nutritional counseling sessions over a period of 2 months.
* Complete assessments that include anthropometric measurements (weight, height, BMI), body composition analysis, and blood tests for total cholesterol, blood glucose, uric acid levels
* Fill out questionnaires to provide information on their attitudes, and health behaviors before and after the intervention.

This study aims to provide insights into the benefits of nutritional counseling in improving various health outcomes among obese female employees.

DETAILED DESCRIPTION:
This quasi-experimental study is conducted over a period of two months and involves 97 obese female employees at Adam Malik Hospital, Medan. The primary aim is to evaluate the effectiveness of nutritional counseling in improving participants' anthropometric measurements, body composition, total cholesterol, blood glucose, uric acid levels, as well as on attitudes, and behavioral changes.

The study design follows a pretest-posttest model with no control group. All participants undergo baseline measurements for anthropometric indicators (weight, height, and BMI), body composition analysis using bioelectrical impedance analysis (BIA), and blood tests for biochemical markers ( total cholesterol, blood glucose, uric acid levels). Nutritional counseling is then provided in sessions where participant receives dietary guidance tailored to their specific needs and health goals.

Data collection also includes demographic information (age, profession, smoking status, alcohol consumption, comorbidities, dietary intake, marital and pregnancy history, socioeconomic status) to offer a broader context for analyzing the outcomes of the intervention. Participants are required to fast for at least 8 hours before blood samples are collected to ensure accurate biochemical assessments.

Upon completion of the counseling intervention, participants will undergo the same assessments as during the pretest phase. The study seeks to detect measurable changes in both behavioral and biological metrics, thereby providing insights into the efficacy of nutritional counseling as a tool for improving health outcomes in an obese working population.

This study also emphasizes the role of structured nutritional education in promoting long-term behavioral change, particularly in settings where employees may face challenges related to weight management. By addressing not only physical health indicators but also psychological factors like knowledge and attitudes, the study aims to contribute to a more holistic approach to workplace health management.

ELIGIBILITY:
Inclusion Criteria:

* Female employees at Adam Malik Hospital, Medan
* Participants aged <65 years
* Participants with a Body Mass Index (BMI) ≥25 kg/m²
* Participants who are willing to follow all stages of the research procedure and sign the informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women with infants under 1 year of age
* Participants undergoing routine treatment with insulin, corticosteroids, antipsychotics, antiepileptics, or beta-blockers
* Participants unable to undergo body composition measurement

Ages: 24 Years to 63 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Weight in Nutritional Counseling | Baseline and 8-week after the intervention
  Weight will be measured using a calibrated body weight scale. Participants will be assessed barefoot, standing upright, and with pockets emptied. Measurements will be recorded to an accuracy of 0.1 kg. Weight will be measured twice: before and after counseling to evaluate changes.
  Outcome Measure: Weight (unit: kg)
Height in Nutritional Counseling | Baseline and 8-week after the intervention
  Height will be measured using a GEA SMIC ZT-120 scale stadiometer. Participants will be assessed barefoot, standing straight with their back, shoulders, buttocks, and heels against the wall. Measurements will be recorded to an accuracy of 0.1 cm. Height will be measured twice: before and after counseling to evaluate changes.
  Outcome Measure: Height (unit: cm)
Body Mass index in Nutritional Counseling | Baseline and 8-week after the intervention
  Body Mass Index (BMI) will be calculated using the formula BMI = weight (kg) / height (m²). Weight will be measured using a calibrated body weight scale and height using a GEA SMIC ZT-120 scale stadiometer. BMI will be calculated after obtaining both measurements, assessed twice: before and after counseling to evaluate changes.
  Outcome Measure: BMI (unit: kg/m²)
Mid-Upper Arm Circumference (MUAC) in Nutritional Counseling | Baseline and 8-week after the intervention
  Mid-Upper Arm Circumference (MUAC) will be measured using the SECA 201 measuring tape. Measurements will be taken at the midpoint between the acromion and olecranon processes of the non-dominant arm, following standard procedures. MUAC will be recorded before and after the nutritional counseling intervention to assess changes in muscle and fat tissue.
Waist Circumference (WC) in Nutritional Counseling | Baseline and 8-week after the intervention
  Waist Circumference (WC) will be measured using the SECA 201 measuring tape at the midpoint between the lowest rib and the iliac crest, following standard anthropometric guidelines. WC measurements will be taken before and after the nutritional counseling intervention to monitor changes in abdominal fat.
Fat Free Mass Index in Nutritional Counseling | Baseline and 8-week after the intervention
  Fat Free Mass Index (FFMI) will be calculated using the formula FFMI = fat free mass (kg) / height (m²). Fat free mass will be assessed using the bioelectrical impedance analysis (BIA) device, SECA 514. Participants will be prepared as per standard guidelines. FFMI will be measured before and after counseling to track changes.
  Outcome Measure: Fat Free Mass Index (unit: kg/m²)
Fat Mass in Nutritional Counseling | Baseline and 8-week after the intervention
  Fat Mass will be calculated using the bioelectrical impedance analysis (BIA) device, SECA 514. Participants will be prepared according to standard guidelines prior to measurement. Fat Mass (in kilograms) will be assessed before and after the nutritional counseling intervention to monitor changes in body composition.
Skeletal Muscle Mass in Nutritional Counseling | Baseline and 8-week after the intervention
  Skeletal Muscle Mass (SMM) will be measured using the bioelectrical impedance analysis (BIA) device, SECA 514. Participants will adhere to standard preparation procedures. SMM will be recorded in kilograms (kg) and assessed before and after counseling to monitor changes.
  Outcome Measure: Skeletal Muscle Mass (unit: kg)
Visceral Adipose Tissue (VAT) in Nutritional Counseling | Baseline and 8-week after the intervention
  Visceral Adipose Tissue (VAT) will be measured using the bioelectrical impedance analysis (BIA) device, SECA 514. Participants will follow standard preparation guidelines before the assessment. VAT will be evaluated before and after the nutritional counseling intervention to monitor changes in visceral fat levels.
Uric Acid Levels in Nutritional Counseling | Baseline and 8-week after the intervention
  Uric acid levels will be measured using the AutoCheck device, a point-of-care testing system. Blood samples will be collected via finger prick without the need for fasting. Measurements will be taken at baseline and 8 weeks after the nutritional counseling intervention to monitor changes in uric acid levels.
  Outcome Measure: Uric Acid (unit: mg/dL or μmol/L)
Blood Glucose Levels in Nutritional Counseling | Baseline and 8-week after the intervention
  Blood glucose levels will be measured using the AutoCheck device, a point-of-care testing system. Blood samples will be collected via finger prick after an overnight fast of at least 8 hours. Measurements will be taken at baseline and 8 weeks after the nutritional counseling intervention to monitor changes in glycemic control.
Total Cholesterol in Nutritional Counseling | Baseline and 8-week after the intervention
  Total cholesterol levels will be measured using the AutoCheck device, a point-of-care testing system. Blood samples will be collected via finger prick after an overnight fast of at least 8 hours. Measurements will be conducted at baseline and 8 weeks after the nutritional counseling intervention to monitor changes in lipid profile.

SECONDARY OUTCOMES:
Attitude in Nutritional Counseling | Baseline and 8 weeks after the intervention
  Attitude will be assessed using a questionnaire adapted from the Weight Self-Stigma Questionnaire (WSSQ) consisting of 12 statements. Participants will respond using a 6-point Likert scale ranging from strongly disagree to strongly agree. Changes in attitude scores will be analyzed to evaluate the effectiveness of the nutritional counseling in modifying participants' attitudes toward weight and eating behaviors.
Behavioral Changes in Nutritional Counseling | Baseline and 8-week after the intervention
  It will be assessed using the Transtheoretical Model (TTM) questionnaire, which consists of two parts: the stages of change and the processes of change. The stages of change section contains 6 statements, and participants select the one statement that best describes their current state. The processes of change section includes 32 items rated on a 5-point Likert scale, measuring participants' engagement in behavioral change processes.

CONTACTS AND LOCATIONS:
Overall Officials: Hilna K Shalihat, Master's, Principal Investigator — Indonesian Association of Clinical Nutrition Specialists
Locations (1):
- Nutrition Unit of Adam Malik Hospital, Medan, North Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to concerns regarding participant confidentiality and lack of appropriate infrastructure to ensure secure data sharing